CLINICAL TRIAL: NCT02660372
Title: A Multi-center, Randomized, Observer-blind, Parallel Group, 8-weeks Non-inferiority Clinical Trial to Compare the Efficacy and Safety of Two Brands of Simeticone for Symptomatic Treatment of Functional Dyspepsia in Adults
Brief Title: Efficacy and Safety of Two Simeticone Brands in Adults With Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO-150121160547-DHCT
Record Dates: First submitted 2016-01-11; First posted 2016-01-21 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Espumisan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imonogas (Experimental): Imonogas 120 mg, 1 capsule three times daily for 8 weeks
  Interventions: Drug: Imonogas
- Espumisan (Active Comparator): Espumisan 40 mg, 2 capsules four times daily for 8 weeks
  Interventions: Drug: Espumisan

INTERVENTIONS:
Drug: Imonogas — Simethicone 120 mg in gel capsules
  Other Names: Imogas
  Arms: Imonogas
Drug: Espumisan — Simethicone 40 mg in gel capsules
  Arms: Espumisan

SUMMARY:
The aim of this study is to show non-inferiority of two brands of simeticone in adult patients suffering from functional dyspepsia.

DETAILED DESCRIPTION:
This is a multi-center, randomized, observer-blind, parallel-group, 8-weeks, non-inferiority clinical trial to compare the efficacy and safety of two brands of Simeticone for symptomatic treatment of functional dyspepsia in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of the age of 18 years or older with a suspected diagnosis of functional dyspepsia according to Rome III criteria (see Appendix A) e.g. subjects suffering from bothersome postprandial fullness or early satiation or epigastric pain or epigastric burning AND no evidence of structural disease (including upper GI endoscopy) that is likely to explain the symptoms. Criteria fulfilled for the last 3 months. Symptom onset at least 6 months prior to diagnosis.
2. Have a Body Mass Index (BMI) between 18.5-30.
3. Absence of significant structural/organic abnormalities on abdominal ultrasound and upper gastrointestinal endoscopy performed within the last 3 months prior to baseline to exclude a structural cause for the symptoms.
4. Negative Helicobacter Pylori urea breath test.
5. Presence of at least three out of the assessed ten symptoms judged to be at least of moderate or severe intensity, assessed after withdrawal of any medication potentially affecting the gastrointestinal tract and at least 7 days wash-out period.
6. Females of childbearing potential must have a negative urine pregnancy test at the baseline visit.
7. Male or non-pregnant, non-lactating female agree to the contraceptive requirements (including female partner's use of a highly effective form of birth control for at least 3 months before the study, during the study and for 3 months after the last dose of study drug) as outlined in Section 10.7.4.
8. Able to read and understand the local language;
9. Provide a signed and dated informed consent form prior to any study-related procedures;
10. Willing and able to comply with all study procedures and attend the scheduled visits for the duration of the study.

Exclusion Criteria:

1. Subjects meeting the diagnostic Rome III criteria for Irritable Bowel Disease (IBS) (see Appendix A).
2. a) severe gastroesophageal reflux symptoms (typical symptoms - heartburn, regurgitation, dysphagia, odynophagia, and/or signs of reflux at upper GI endoscopy) at Screening visit.

   b) predominant gastroesophageal reflux symptoms defined as a Subject's Symptom Severity Score of 2 or more for heartburn and regurgitation at Baseline visit after the 7-days wash-out period (see questionnaire in Appendix B).
3. Significant medical condition which may interfere with a subject's participation in the study, e.g. diabetes mellitus, thyroid dysfunction, renal insufficiency, congestive heart failure, electrolyte disturbances or autoimmune diseases requiring immunosuppressive treatment.
4. Known hepatic, biliary or pancreatic disease.
5. Known lactose or gluten intolerance or celiac disease.
6. Known HIV positive or AIDS.
7. Suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates).
8. Unwillingness or inability to withdraw and abstain from medication which is likely to affect gastrointestinal function or symptoms during the 7-days wash-out period and throughout the study period, including the following drugs:

   * gastrointestinal medications including antispasmodics, prokinetics, proton pump inhibitors, H2 blockers, antacids, alginate, bismuth preparations, sucralfate, misoprostol, charcoal, diosmectite, enzymes (e.g. Kreon®, Mezim®).
   * other medications that could interfere with gastrointestinal function e.g. antibiotics (except for local application), theophylline, NSAIDs (except for low-dose aspirin for prevention of heart disease), opioid analgesics, codeine, ulcerogenic substances (e.g. oral glucocorticoids), anxiolytics, neuroleptics, antidepressants, and/or others in the judgment of the investigator.
9. Females who are pregnant or breastfeeding.
10. Males with a pregnant partner or a partner who is currently trying to become pregnant.
11. Known sensitivity to the investigational products.
12. Subjects who were previously screened and ineligible or were randomized to receive investigational product.
13. Currently participating in another clinical trial or has done so in the past 30 days.
14. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., principal investigator, subinvestigators, study coordinators, other site personnel, employees of Johnson & Johnson LLC or McNeil AB subsidiaries, contractors of Johnson & Johnson LLC or McNeil AB, and the families of each).
15. Other severe, acute or chronic, medical or psychiatric condition(s) or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Aggregate symptom score calculated from subjects assessment of 10 individual upper gastrointestinal symptoms 8 weeks after start of treatments | 8 weeks
  Specific questionnaire with a 4 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, Study Director — McNeil AB
Locations (1):
- City Polyclinic #2 of Moscow Health Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided